CLINICAL TRIAL: NCT01481597
Title: Tolerance and Pharmacokinetics of Single-dose Intravenous Deuteporfin in Healthy Volunteers
Brief Title: Deuteporfin Tolerance and Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDZJ1109DT
Record Dates: First submitted 2011-10-10; First posted 2011-11-29 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: deuteporfin; safety; tolerability; pharmacokinetics; healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- deuteporfin 1mg/kg (Experimental)
  Interventions: Drug: deuteporfin
- deuteporfin 2.5mg/kg (Active Comparator)
  Interventions: Drug: deuteporfin
- deuteporfin 5mg/kg (Active Comparator)
  Interventions: Drug: deuteporfin
- deuteporfin 7.5mg/kg (Active Comparator)
  Interventions: Drug: deuteporfin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: deuteporfin — deuteporfin 1 mg/kg IV as a single dose
  Arms: deuteporfin 1mg/kg
Drug: deuteporfin — deuteporfin 2.5 mg/kg IV as a single dose
  Arms: deuteporfin 2.5mg/kg
Drug: deuteporfin — deuteporfin 5 mg/kg IV as a single dose
  Arms: deuteporfin 5mg/kg
Drug: deuteporfin — deuteporfin 7.5 mg/kg IV as a single dose
  Arms: deuteporfin 7.5mg/kg
Drug: placebo — Placebo for 2.5 mg/kg, 5 mg/kg and 7.5mg/kg of deuteporfin (single dose)
  Arms: placebo

SUMMARY:
Deuteporfin, a novel photodynamic drug developed in China, displays good photodynamic antitumor activity. The purpose of the present study is to investigate the safety and pharmacokinetics of intravenous deuteporfin in healthy Chinese volunteers following single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male and/or female subjects
* 18 to 45 years old with Body mass index (BMI) within the range of 19 to 24 kg/m2
* weigh at least 45 kg for female subjects or 50 kg for male subjects
* In good health as confirmed by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis on the screening and baseline evaluation
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Significant illness or major surgery within four weeks prior to dosing
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies and photoallergy)
* Use of any drugs which might interfere with drug absorption, distribution, metabolism, excretion or cause photoallergy within 30 days prior to dosing, or any drugs within 14 days prior to dosing
* Participation in any clinical investigation within 30 days prior to dosing
* Smokers, alcoholics, drug abusers
* Immunodeficiency diseases, including a positive HIV test result, Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result
* pregnancy or lactation for female subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
number of participants with adverse events | up to 19 days following injection
  number of participants with adverse events as a measure of safety and tolerability of single dose of deuteporfin administered to healthy subjects

SECONDARY OUTCOMES:
Pharmacokinetic profile | predose, 20, 40 and 60 min during-dose, and 5, 10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8 ,12, 24h post-dose
  Pharmacokinetic profile: Cmax (Peak Concentration), AUC (area under the plasma-concentration-time curve ), T1/2 (half life)

CONTACTS AND LOCATIONS:
Overall Officials: Zeneng Cheng, Ph.D, Principal Investigator — Xiangya Hospital of Central South University; Jining Tao, Master, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.; Pingsheng Xu, Master, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central-South University, Changsha, Hunan, China